CLINICAL TRIAL: NCT06445985
Title: Hydrotherapy for Health in Boys and Adolescents With Duchenne Muscular Dystrophy
Brief Title: Hydrotherapy in Duchenne Muscular Dystrophy (DMD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Duchenne UK (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 304633; 21/PR/1748 (Other: Health Research Authority)
Record Dates: First submitted 2024-02-14; First posted 2024-06-06 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Patients with DMD, show great variability in age and speed of deterioration. As such it is difficult to find matched controls for a short randomised intervention study. Instead, due to the progressive nature of DMD and the inherent variance within a mixed age and ability population, the participants will act as their own controls. This single-arm, non-crossover design where the participant acts as his own control, although not as robust as randomized control exercise trials, is advocated for longitudinal interventions in populations such as the present one.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will have a 12 week period where they will continue with their habitual physical activity behaviour. Diet and physical activity will be monitored
- Hydrotherapy (Active Comparator): Participants will complete 12-weeks of hydrotherapy, involving up to 60 mins of hydrotherapy once a week. Diet and physical activity will be monitored.
  Interventions: Other: Hydrotherapy

INTERVENTIONS:
Other: Hydrotherapy — Physiotherapy led pool session
  Arms: Hydrotherapy

SUMMARY:
The goal of this clinical trial aims to establish if there are meaningful benefits to providing a hydrotherapy service for young people with Duchenne muscular dystrophy (DMD). The main aims are to: 1. to allocate a clinical physiotherapist to a project implementing hydrotherapy in young patients with DMD to establish whether there are meaningful benefits to their daily life. 2. to conduct patient and parent interviews to understand the barriers to completing a hydrotherapy intervention and ensure future research addresses meaningful outcomes for those with DMD.

DETAILED DESCRIPTION:
The quality of life in young males with Duchenne muscular dystrophy (DMD) is negatively impacted by daily pain, changes in body composition and a lack of support to undertake physical activity. Hydrotherapy represents a potential means of involving boys and adolescents with DMD in activity that could benefit the negative factors influencing their quality of life. There are presently no guidelines or evidence for the benefits of hydrotherapy with the standards of care for young males with DMD.

This trial will provide evidence that will allow care providers to advocate the use of hydrotherapy within the management of DMD, as an inclusive activity, that can be adopted by those with DMD who are either ambulatory, or non-ambulatory. Through 12-weeks of hydrotherapy, the trial will investigate whether there are benefits to physical function, pain and quality of life. These measures represent meaningful outcomes in the progression of DMD, and have direct patient impact for those affected by DMD. On completion of the hydrotherapy, there will be a series of interviews with some of the participants and their parents. The aim of these interviews is to understand participant and parent barriers to hydrotherapy, and uncover whether hydrotherapy improves the lives of the participants beyond simple clinical measures and questionnaires.

The study aims recruit 44 boys and young men with Duchenne muscular dystrophy. Patients will be recruited from NHS neuromuscular services and through families who attend the local hospice.

Following an informed consent process they will enter the first 12 week stage, as a control to observe and measure their habitual physical activity, along with monitoring their diet. They will then enter the intervention stage where they will have a weekly physiotherapy led pool session with a number of physical activities. During the hydrotherapy period, participants will access the hydrotherapy pool once a week for 12 weeks. Sessions are supervised by an experienced physiotherapist, who will guide the exercise for a session lasting 30 to 60 minutes.

The exercises, intensity and specific hydrotherapy plan will be derived from consultation with the participants and their parents. Due to the variance within the presentation of the condition, and the inclusive age range within the study, an externally valid approach to exercise prescription will be utilised. Diet and physical function will be measured during this stage.

There will be a number of assessments to be completed at 3 time points. As much as possible these will be arranged as single visits. The first before the control period, the second after the control period, and the third after the hydrotherapy period. The assessments include a number of physical assessments, including assessments of function and ability, body mass and quality of life. After completion, all participants will be invited to complete a qualitative interview, in particular enquiring about the experience and logistics of hydrotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Duchenne Muscular Dystrophy (either by genetics or muscle biopsy)
* Between 6 and 25 years of age
* On stable dose of steroids or not on steroids

Exclusion Criteria:

* Younger than 6 years, older than 25 years
* Recent change in steroid dose, less than 3 months prior
* Undertaking formal hydrotherapy supervised by physiotherapist on a regular basis (weekly or more frequent)

Ages: 6 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — DMD affects those born male.
Enrollment: 31 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass via Bioelectrical impedance (BIA) | 24 weeks
  Fat mass, body fat percentage and fat free mass will be measured using BIA (bioelectrical impedance). BIA has been validated in DMD and is accurate enough to measure longitudinal changes in body composition and muscle mass in this population
Pain Scale | 24 weeks
  A pain map assessment of the topographic distribution of daily pain will also be competed, consistent with our previous work in DMD. Scale of 1-10
PedsQL QoL / DMD QoL - Quality of Life | 24 weeks
  PedsQL QoL - Quality of Life for both participants, and the DMD-QoL Proxy for parents - Scale of 0-4

SECONDARY OUTCOMES:
Upper Limb Strength | 24 weeks
  Upper limb strength using grip and pinch measure using digital, handheld dynamometers North-Star
Range of Motion | 24 weeks
  Limited ankle range of motion (ROM) Ankle plantarflexion-dorsiflexion (PF-DF ROM) will be assessed through a goniometer
Pulmonary function | 24 weeks
  Pulmonary function will be assessed using digital spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Goede, Principal Investigator — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (1):
- Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results of this study will be used to inform the neuromuscular service in Preston and at other sites in the UK. The results will also be shared more widely by presenting them at regional and or national meetings. The results may be published in a scientific journal and presented at scientific medical conferences and through publications and meetings organised by Duchenne UK.

DOCUMENTS (1):
  • Study Protocol (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT06445985/Prot_000.pdf